CLINICAL TRIAL: NCT02712320
Title: An Open-Label, Single-Arm Study of the Safety, Efficacy, and Pharmacokinetic Behavior of Leuprolide Mesylate for Injectable Suspension (LMIS 50 mg) in Subjects With Advanced Prostate Carcinoma - SAFETY EXTENSION
Brief Title: Open-Label Safety Extension Study in Patients Who Have Previously Participated and Have Benefited From LMIS 50 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS-Qualitix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP01C-13-001-EX
Record Dates: First submitted 2016-02-22; First posted 2016-03-18 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Neoplasm Cancer Carcinoma; Safety Extension
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LMIS 50 mg (Experimental): 50 mg leuprolide mesylate administered subcutaneously, when given as two separate injections 6 months apart (Month 12 and Month 18 from the initiation of Protocol FP01C-13-001)
  Interventions: Drug: LMIS 50 mg

INTERVENTIONS:
Drug: LMIS 50 mg — Subcutaneous injection of 50 mg Leuprolide Mesylate

SUMMARY:
This is a safety extension of up to 12 months of additional treatment with LMIS 50 mg after the subject has completed 12 months of treatment under Protocol FP01C-13-001 and remain eligible for continued treatment with androgen deprivation therapy. Subjects participating in Protocol FP01C-13-001-EX will be followed for safety only.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single-arm safety extension study. After completing 12 months of treatment with LMIS 50 mg under Protocol FP01C-13-001 (with last dose under Protocol FP01C-13-001 approximately 6 months prior to Day 0 or Protocol FP01C-13-001-EX) and providing a written informed consent, subjects will be screened against baseline inclusion/exclusion criteria necessary for study eligibility. Eligible subjects will receive LMIS 50 mg from the prefilled syringes (without dilution or other mixing) in up to two single subcutaneous injections given 6 months apart.

ELIGIBILITY:
Inclusion Criteria:

1. Complete 12 months of treatment with LMIS 50 mg under Protocol FP01C-13-001. If a subject wishes to enter the Extension study after more than 28 days following his end of study visit for Protocol FP01C-13-001, his serum testosterone level should be repeated at the screening visit to confirm that his castrate-level testosterone has been maintained.
2. Laboratory values

   * Absolute neutrophil count ≥ 1,500 cells/µL
   * Platelets≥100,000 cells/µL
   * Hemoglobin ≥ 10 gm/dL
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Aspartate Transaminase (AST/SGOT) ≤ 2.5 × ULN
   * Alanine Aminotransferase (ALT/SGPT) ≤ 2.5 × ULN
   * Serum creatinine ≤ 1.5 mg/dL
   * Lipid profile within acceptable range according to investigator's opinion
   * Serum glucose within acceptable range according to investigator's opinion
   * HgbA1c within acceptable range according to investigator's opinion
   * Clinical chemistries (K, Na, Mg, Ca and P) within acceptable range according to investigator's judgment
   * Urinalysis within normal range according to the investigator's judgment
3. Agree to use male contraceptive methods during study trial
4. In the Investigator's opinion, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol
5. All aspects of the protocol explained and written informed consent obtained *If the patient completed 12 months of treatment with LMIS 50 mg more than 28 days prior to entering the Extension study, the Eastern Cooperative Oncology Group (ECOG), Physical Examination (PE), ECG, laboratory and Prostate Specific Antigen (PSA) tests should be repeated.

If the patient has completed 12 months of treatment with LMIS 50 mg under Protocol FP01C-13-001 within the last 28 days, they will be allowed to enter the Extension study without repeating the testosterone measurements, ECG, PE, laboratory and the PSA tests

Exclusion Criteria:

1. Receipt of chemotherapy, immunotherapy, cryotherapy, radiotherapy, or anti-androgen therapy other than LMIS 50 mg under Protocol FP01C-13-001 for treatment of carcinoma of the prostate during the subject's participation in Protocol FP01C-13-001. Radiation for pain control will be allowed during the study.
2. Receipt of any Luteinizing Hormone-releasing Hormone (LHRH) suppressive therapy within 6 months of Screening Visit other than LMIS 50 mg under Protocol FP01C-13-001
3. Subject has used prohibited treatments as listed in the Section 8.2 during participation in Protocol FP01C-13-001.
4. Any pathological event, clinical adverse event, or any change in the subject's status at the end of FP01C-13-001 giving indication to the investigator that further participation in the study may not be the best interest of the subject
5. Investigator considers that it is no longer feasible for the subject to be included in a study of LMIS 50 mg
6. Subjects with persistent, non-castrate testosterone levels judged by the investigator
7. Uncontrolled intercurrent illness that would jeopardize the subject's safety, interfere with the objectives of the protocol, or limit the subject's compliance with study requirements, as determined by the Investigator in consultation with the Sponsor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mao, Ph.D., Study Director — Foresee Pharmaceuticals Co., Ltd.
Locations (7):
- United States (7):
  - Urology Centers of Alabama, Homewood, Alabama
  - Genesis Research, LLC, San Diego, California
  - Idaho Urologic Institute - Meridian, Meridian, Idaho
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Carolina Clinical Trials, LLC, Concord, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Seattle Urology Research Center, Burien, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were males with advanced prostate carcinoma that completed 12 months (48-week) of therapy with Leuprolide Mesylate Injectable Suspension (LMIS) 50 mg under the Protocol FP01C-13-001 and were suitable candidates for continued medical androgen ablation therapy as judged by investigators.
Groups:
- LMIS 50 mg: All subjects were males with advanced prostate carcinoma. They were injected 2 doses of LMIS 50 mg with approximately 6 months (24-week) apart (Month 12 and Month 18 from the initiation of Protocol FP01C-13-001)
  LMIS 50 mg: Subcutaneous injection of 50 mg Leuprolide Mesylate
Period: Overall Study
Arm/Group | LMIS 50 mg
Started | 30
Completed | 25
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Transferred to another facility | 1
Not completed — Treating with the prohibited medications | 2

BASELINE CHARACTERISTICS:
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Evaluate the incidence of adverse events, drug-related adverse events, and serious adverse events
Time Frame: Up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Participants
  TEAE | 12
  Drug-related AE | 1
  Serious Adverse Event (SAE) | 4

2. Primary Outcome: Evaluate the Effect of LMIS 50 mg on Cardiovascular Function
Description: Use 12-lead resting electrocardiograms (ECGs) to evaluate the effect of LMIS 50 mg on cardiovascular function, such as heart rate, RR interval, QRS complex, PR interval, and QT interval.
Time Frame: Up to 48 weeks
Population: 8 subjects did not receive the second dose due to drug supply expiration, and 4 subjects due to early termination. Hence, only 18 subjects entered Day 168 (V4). 3 subjects were unable or unwilling to return on Day 336 (V6/EOS) due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Participants
  Overall Interpretation at Screening (V1): number analyzed (Participants) | 29
  Overall Interpretation at Screening (V1): Normal | 4
  Overall Interpretation at Screening (V1): Abnormal-No clinical significance | 25
  Overall Interpretation on Day 168 (V4): number analyzed (Participants) | 18
  Overall Interpretation on Day 168 (V4): Normal | 2
  Overall Interpretation on Day 168 (V4): Abnormal-No clinical significance | 16
  Overall Interpretation on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Overall Interpretation on Day 336 (V6/EOS): Normal | 7
  Overall Interpretation on Day 336 (V6/EOS): Abnormal-No clinical significance | 20

3. Primary Outcome: Laboratory Assessments - Hematology
Description: Hematology assessments performed in this study included hemoglobin, hematocrit, Red Blood Cell (RBC), White Blood Cell (WBC), platelets, neutrophil, eosinophil, basophil, lymphocyte, monocyte, and HbA1c.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Participants
  Hemoglobin (gm/dL) at Screening (V1): Normal | 17
  Hemoglobin (gm/dL) at Screening (V1): Abnormal-No clinical significance | 13
  Hemoglobin (gm/dL) at Screening (V1): Abnormal-Clinical significance | 0
  Hemoglobin (gm/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Hemoglobin (gm/dL) on Day 168 (V4): Normal | 9
  Hemoglobin (gm/dL) on Day 168 (V4): Abnormal-No clinical significance | 9
  Hemoglobin (gm/dL) on Day 168 (V4): Abnormal-Clinical significance | 0
  Hemoglobin (gm/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Hemoglobin (gm/dL) on Day 336 (V6/EOS): Normal | 13
  Hemoglobin (gm/dL) on Day 336 (V6/EOS): Abnormal-No clinical significance | 14
  Hemoglobin (gm/dL) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Hematocrit (%) at Screening (V1): Normal | 18
  Hematocrit (%) at Screening (V1): Abnormal-No clinical significance | 12
  Hematocrit (%) at Screening (V1): Abnormal-Clinical significance | 0
  Hematocrit (%) on Day 168 (V4): number analyzed (Participants) | 18
  Hematocrit (%) on Day 168 (V4): Normal | 4
  Hematocrit (%) on Day 168 (V4): Abnormal-No clinical significance | 14
  Hematocrit (%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Hematocrit (%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Hematocrit (%) on Day 336 (V6/EOS): Normal | 7
  Hematocrit (%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 20
  Hematocrit (%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  RBC (x10.e6/uL) at Screening (V1): Normal | 15
  RBC (x10.e6/uL) at Screening (V1): Abnormal-No clinical significance | 15
  RBC (x10.e6/uL) at Screening (V1): Abnormal-Clinical significance | 0
  RBC (x10.e6/uL) on Day 168 (V4): number analyzed (Participants) | 18
  RBC (x10.e6/uL) on Day 168 (V4): Normal | 2
  RBC (x10.e6/uL) on Day 168 (V4): Abnormal-No clinical significance | 16
  RBC (x10.e6/uL) on Day 168 (V4): Abnormal-Clinical significance | 0
  RBC (x10.e6/uL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  RBC (x10.e6/uL) on Day 336 (V6/EOS): Normal | 6
  RBC (x10.e6/uL) on Day 336 (V6/EOS): Abnormal-No clinical significance | 21
  RBC (x10.e6/uL) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  WBC (x10.e3/uL) at Screening (V1): Normal | 26
  WBC (x10.e3/uL) at Screening (V1): Abnormal-No clinical significance | 4
  WBC (x10.e3/uL) at Screening (V1): Abnormal-Clinical significance | 0
  WBC (x10.e3/uL) on Day 168 (V4): number analyzed (Participants) | 18
  WBC (x10.e3/uL) on Day 168 (V4): Normal | 18
  WBC (x10.e3/uL) on Day 168 (V4): Abnormal-No clinical significance | 0
  WBC (x10.e3/uL) on Day 168 (V4): Abnormal-Clinical significance | 0
  WBC (x10.e3/uL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  WBC (x10.e3/uL) on Day 336 (V6/EOS): Normal | 22
  WBC (x10.e3/uL) on Day 336 (V6/EOS): Abnormal-No clinical significance | 5
  WBC (x10.e3/uL) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Platelets (x10.e3/uL) at Screening (V1): Normal | 27
  Platelets (x10.e3/uL) at Screening (V1): Abnormal-No clinical significance | 3
  Platelets (x10.e3/uL) at Screening (V1): Abnormal-Clinical significance | 0
  Platelets (x10.e3/uL) on Day 168 (V4): number analyzed (Participants) | 18
  Platelets (x10.e3/uL) on Day 168 (V4): Normal | 14
  Platelets (x10.e3/uL) on Day 168 (V4): Abnormal-No clinical significance | 4
  Platelets (x10.e3/uL) on Day 168 (V4): Abnormal-Clinical significance | 0
  Platelets (x10.e3/uL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Platelets (x10.e3/uL) on Day 336 (V6/EOS): Normal | 23
  Platelets (x10.e3/uL) on Day 336 (V6/EOS): Abnormal-No clinical significance | 4
  Platelets (x10.e3/uL) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Neutrophils(%) at Screening (V1): Normal | 28
  Neutrophils(%) at Screening (V1): Abnormal-No clinical significance | 2
  Neutrophils(%) at Screening (V1): Abnormal-Clinical significance | 0
  Neutrophils(%) on Day 168 (V4): number analyzed (Participants) | 17
  Neutrophils(%) on Day 168 (V4): Normal | 15
  Neutrophils(%) on Day 168 (V4): Abnormal-No clinical significance | 2
  Neutrophils(%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Neutrophils(%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Neutrophils(%) on Day 336 (V6/EOS): Normal | 22
  Neutrophils(%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 4
  Neutrophils(%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 1
  Eosinophils(%) at Screening (V1): Normal | 25
  Eosinophils(%) at Screening (V1): Abnormal-No clinical significance | 5
  Eosinophils(%) at Screening (V1): Abnormal-Clinical significance | 0
  Eosinophils(%) on Day 168 (V4): number analyzed (Participants) | 17
  Eosinophils(%) on Day 168 (V4): Normal | 15
  Eosinophils(%) on Day 168 (V4): Abnormal-No clinical significance | 2
  Eosinophils(%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Eosinophils(%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Eosinophils(%) on Day 336 (V6/EOS): Normal | 20
  Eosinophils(%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 7
  Eosinophils(%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Basophils (%) at Screening (V1): Normal | 30
  Basophils (%) at Screening (V1): Abnormal-No clinical significance | 0
  Basophils (%) at Screening (V1): Abnormal-Clinical significance | 0
  Basophils (%) on Day 168 (V4): number analyzed (Participants) | 17
  Basophils (%) on Day 168 (V4): Normal | 16
  Basophils (%) on Day 168 (V4): Abnormal-No clinical significance | 1
  Basophils (%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Basophils (%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Basophils (%) on Day 336 (V6/EOS): Normal | 27
  Basophils (%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 0
  Basophils (%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Lymphocytes (%) at Screening (V1): Normal | 28
  Lymphocytes (%) at Screening (V1): Abnormal-No clinical significance | 2
  Lymphocytes (%) at Screening (V1): Abnormal-Clinical significance | 0
  Lymphocytes (%) on Day 168 (V4): number analyzed (Participants) | 17
  Lymphocytes (%) on Day 168 (V4): Normal | 14
  Lymphocytes (%) on Day 168 (V4): Abnormal-No clinical significance | 3
  Lymphocytes (%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Lymphocytes (%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Lymphocytes (%) on Day 336 (V6/EOS): Normal | 21
  Lymphocytes (%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 6
  Lymphocytes (%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  Monocytes (%) at Screening (V1): Normal | 26
  Monocytes (%) at Screening (V1): Abnormal-No clinical significance | 4
  Monocytes (%) at Screening (V1): Abnormal-Clinical significance | 0
  Monocytes (%) on Day 168 (V4): number analyzed (Participants) | 17
  Monocytes (%) on Day 168 (V4): Normal | 15
  Monocytes (%) on Day 168 (V4): Abnormal-No clinical significance | 2
  Monocytes (%) on Day 168 (V4): Abnormal-Clinical significance | 0
  Monocytes (%) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Monocytes (%) on Day 336 (V6/EOS): Normal | 24
  Monocytes (%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 3
  Monocytes (%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0
  HgbA1c (%) at Screening (V1): Normal | 22
  HgbA1c (%) at Screening (V1): Abnormal-No clinical significance | 8
  HgbA1c (%) at Screening (V1): Abnormal-Clinical significance | 0
  HgbA1c (%) on Day 336 (V6/EOS): number analyzed (Participants) | 24
  HgbA1c (%) on Day 336 (V6/EOS): Normal | 14
  HgbA1c (%) on Day 336 (V6/EOS): Abnormal-No clinical significance | 10
  HgbA1c (%) on Day 336 (V6/EOS): Abnormal-Clinical significance | 0

4. Primary Outcome: Laboratory Assessments - Biochemistry
Description: Biochemical assessments performed in this study included Alanine Aminotransferase (ALT), Aspartate Transaminase (AST), Alkaline Phosphatase (ALP), total bilirubin, Blood Urea Nitrogen (BUN), serum Cr, potassium, sodium, magnesium, calcium, phosphorus, blood glucose, Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), and triglycerides.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Participants
  ALT (U/L) at Screening (V1): Normal | 28
  ALT (U/L) at Screening (V1): Abnormal - No clinical significance | 2
  ALT (U/L) at Screening (V1): Abnormal - Clinical significance | 0
  ALT (U/L) on Day 168 (V4): number analyzed (Participants) | 18
  ALT (U/L) on Day 168 (V4): Normal | 17
  ALT (U/L) on Day 168 (V4): Abnormal - No clinical significance | 1
  ALT (U/L) on Day 168 (V4): Abnormal - Clinical significance | 0
  ALT (U/L) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  ALT (U/L) on Day 336 (V6/EOS): Normal | 26
  ALT (U/L) on Day 336 (V6/EOS): Abnormal - No clinical significance | 1
  ALT (U/L) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  AST (U/L) at Screening (V1): Normal | 29
  AST (U/L) at Screening (V1): Abnormal - No clinical significance | 1
  AST (U/L) at Screening (V1): Abnormal - Clinical significance | 0
  AST (U/L) on Day 168 (V4): number analyzed (Participants) | 18
  AST (U/L) on Day 168 (V4): Normal | 16
  AST (U/L) on Day 168 (V4): Abnormal - No clinical significance | 2
  AST (U/L) on Day 168 (V4): Abnormal - Clinical significance | 0
  AST (U/L) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  AST (U/L) on Day 336 (V6/EOS): Normal | 25
  AST (U/L) on Day 336 (V6/EOS): Abnormal - No clinical significance | 2
  AST (U/L) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  ALP (U/L) at Screening (V1): Normal | 26
  ALP (U/L) at Screening (V1): Abnormal - No clinical significance | 3
  ALP (U/L) at Screening (V1): Abnormal - Clinical significance | 1
  ALP (U/L) on Day 168 (V4): number analyzed (Participants) | 18
  ALP (U/L) on Day 168 (V4): Normal | 10
  ALP (U/L) on Day 168 (V4): Abnormal - No clinical significance | 8
  ALP (U/L) on Day 168 (V4): Abnormal - Clinical significance | 0
  ALP (U/L) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  ALP (U/L) on Day 336 (V6/EOS): Normal | 17
  ALP (U/L) on Day 336 (V6/EOS): Abnormal - No clinical significance | 10
  ALP (U/L) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Total bilirubin(mg/dL) at Screening (V1): Normal | 30
  Total bilirubin(mg/dL) at Screening (V1): Abnormal - No clinical significance | 0
  Total bilirubin(mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Total bilirubin(mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Total bilirubin(mg/dL) on Day 168 (V4): Normal | 18
  Total bilirubin(mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 0
  Total bilirubin(mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Total bilirubin(mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Total bilirubin(mg/dL) on Day 336 (V6/EOS): Normal | 27
  Total bilirubin(mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 0
  Total bilirubin(mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  BUN (mg/dL) at Screening (V1): Normal | 21
  BUN (mg/dL) at Screening (V1): Abnormal - No clinical significance | 9
  BUN (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  BUN (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  BUN (mg/dL) on Day 168 (V4): Normal | 9
  BUN (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 9
  BUN (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  BUN (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  BUN (mg/dL) on Day 336 (V6/EOS): Normal | 15
  BUN (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 12
  BUN (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Serum Cr. (mg/dL) at Screening (V1): Normal | 27
  Serum Cr. (mg/dL) at Screening (V1): Abnormal - No clinical significance | 3
  Serum Cr. (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Serum Cr. (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Serum Cr. (mg/dL) on Day 168 (V4): Normal | 15
  Serum Cr. (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 3
  Serum Cr. (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Serum Cr. (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Serum Cr. (mg/dL) on Day 336 (V6/EOS): Normal | 24
  Serum Cr. (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 3
  Serum Cr. (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Potassium (mEq/L) at Screening (V1): Normal | 28
  Potassium (mEq/L) at Screening (V1): Abnormal - No clinical significance | 2
  Potassium (mEq/L) at Screening (V1): Abnormal - Clinical significance | 0
  Potassium (mEq/L) on Day 168 (V4): number analyzed (Participants) | 18
  Potassium (mEq/L) on Day 168 (V4): Normal | 18
  Potassium (mEq/L) on Day 168 (V4): Abnormal - No clinical significance | 0
  Potassium (mEq/L) on Day 168 (V4): Abnormal - Clinical significance | 0
  Potassium (mEq/L) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Potassium (mEq/L) on Day 336 (V6/EOS): Normal | 26
  Potassium (mEq/L) on Day 336 (V6/EOS): Abnormal - No clinical significance | 1
  Potassium (mEq/L) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Sodium (mEq/L) at Screening (V1): Normal | 30
  Sodium (mEq/L) at Screening (V1): Abnormal - No clinical significance | 0
  Sodium (mEq/L) at Screening (V1): Abnormal - Clinical significance | 0
  Sodium (mEq/L) on Day 168 (V4): number analyzed (Participants) | 18
  Sodium (mEq/L) on Day 168 (V4): Normal | 17
  Sodium (mEq/L) on Day 168 (V4): Abnormal - No clinical significance | 1
  Sodium (mEq/L) on Day 168 (V4): Abnormal - Clinical significance | 0
  Sodium (mEq/L) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Sodium (mEq/L) on Day 336 (V6/EOS): Normal | 26
  Sodium (mEq/L) on Day 336 (V6/EOS): Abnormal - No clinical significance | 1
  Sodium (mEq/L) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Magnesium (mg/dL) at Screening (V1): Normal | 26
  Magnesium (mg/dL) at Screening (V1): Abnormal - No clinical significance | 4
  Magnesium (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Magnesium (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Magnesium (mg/dL) on Day 168 (V4): Normal | 14
  Magnesium (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 4
  Magnesium (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Magnesium (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Magnesium (mg/dL) on Day 336 (V6/EOS): Normal | 23
  Magnesium (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 4
  Magnesium (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Calcium (mg/dL) at Screening (V1): Normal | 29
  Calcium (mg/dL) at Screening (V1): Abnormal - No clinical significance | 1
  Calcium (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Calcium (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Calcium (mg/dL) on Day 168 (V4): Normal | 17
  Calcium (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 1
  Calcium (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Calcium (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Calcium (mg/dL) on Day 336 (V6/EOS): Normal | 25
  Calcium (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 2
  Calcium (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Phosphorus (mg/dL) at Screening (V1): Normal | 29
  Phosphorus (mg/dL) at Screening (V1): Abnormal - No clinical significance | 1
  Phosphorus (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Phosphorus (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Phosphorus (mg/dL) on Day 168 (V4): Normal | 16
  Phosphorus (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 2
  Phosphorus (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Phosphorus (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Phosphorus (mg/dL) on Day 336 (V6/EOS): Normal | 25
  Phosphorus (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 2
  Phosphorus (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Blood glucose (mg/dL) at Screening (V1): Normal | 22
  Blood glucose (mg/dL) at Screening (V1): Abnormal - No clinical significance | 8
  Blood glucose (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Blood glucose (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Blood glucose (mg/dL) on Day 168 (V4): Normal | 13
  Blood glucose (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 5
  Blood glucose (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Blood glucose (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Blood glucose (mg/dL) on Day 336 (V6/EOS): Normal | 14
  Blood glucose (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 12
  Blood glucose (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 1
  LDL (mg/dL) at Screening (V1): number analyzed (Participants) | 29
  LDL (mg/dL) at Screening (V1): Normal | 28
  LDL (mg/dL) at Screening (V1): Abnormal - No clinical significance | 1
  LDL (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  LDL (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  LDL (mg/dL) on Day 168 (V4): Normal | 13
  LDL (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 5
  LDL (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  LDL (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 26
  LDL (mg/dL) on Day 336 (V6/EOS): Normal | 19
  LDL (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 7
  LDL (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  HDL (mg/dL) at Screening (V1): Normal | 21
  HDL (mg/dL) at Screening (V1): Abnormal - No clinical significance | 9
  HDL (mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  HDL (mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  HDL (mg/dL) on Day 168 (V4): Normal | 12
  HDL (mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 6
  HDL (mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  HDL (mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  HDL (mg/dL) on Day 336 (V6/EOS): Normal | 21
  HDL (mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 6
  HDL (mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0
  Triglycerides(mg/dL) at Screening (V1): Normal | 17
  Triglycerides(mg/dL) at Screening (V1): Abnormal - No clinical significance | 13
  Triglycerides(mg/dL) at Screening (V1): Abnormal - Clinical significance | 0
  Triglycerides(mg/dL) on Day 168 (V4): number analyzed (Participants) | 18
  Triglycerides(mg/dL) on Day 168 (V4): Normal | 6
  Triglycerides(mg/dL) on Day 168 (V4): Abnormal - No clinical significance | 12
  Triglycerides(mg/dL) on Day 168 (V4): Abnormal - Clinical significance | 0
  Triglycerides(mg/dL) on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Triglycerides(mg/dL) on Day 336 (V6/EOS): Normal | 13
  Triglycerides(mg/dL) on Day 336 (V6/EOS): Abnormal - No clinical significance | 14
  Triglycerides(mg/dL) on Day 336 (V6/EOS): Abnormal - Clinical significance | 0

5. Primary Outcome: Laboratory Assessments - Urinalysis
Description: Urinalysis was performed to assess the safety profile of LMIS 50 mg during the study period, including pH, specific gravity, and the presences of leukocytes, erythrocytes, or protein.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LMIS 50 mg
Number analyzed (Participants) | 30
Participants
  pH at Screening (V1): Normal | 30
  pH at Screening (V1): Abnormal - No clinical significance | 0
  pH on Day 168 (V4): number analyzed (Participants) | 18
  pH on Day 168 (V4): Normal | 18
  pH on Day 168 (V4): Abnormal - No clinical significance | 0
  pH on Day 336 (V6/EOS): number analyzed (Participants) | 27
  pH on Day 336 (V6/EOS): Normal | 27
  pH on Day 336 (V6/EOS): Abnormal - No clinical significance | 0
  Specific gravity at Screening (V1): Normal | 30
  Specific gravity at Screening (V1): Abnormal - No clinical significance | 0
  Specific gravity on Day 168 (V4): number analyzed (Participants) | 18
  Specific gravity on Day 168 (V4): Normal | 18
  Specific gravity on Day 168 (V4): Abnormal - No clinical significance | 0
  Specific gravity on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Specific gravity on Day 336 (V6/EOS): Normal | 26
  Specific gravity on Day 336 (V6/EOS): Abnormal - No clinical significance | 1
  Leukocyte at Screening (V1): Normal | 27
  Leukocyte at Screening (V1): Abnormal - No clinical significance | 3
  Leukocyte on Day 168 (V4): number analyzed (Participants) | 18
  Leukocyte on Day 168 (V4): Normal | 16
  Leukocyte on Day 168 (V4): Abnormal - No clinical significance | 2
  Leukocyte on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Leukocyte on Day 336 (V6/EOS): Normal | 23
  Leukocyte on Day 336 (V6/EOS): Abnormal - No clinical significance | 4
  Erythrocyte at Screening (V1): Normal | 28
  Erythrocyte at Screening (V1): Abnormal - No clinical significance | 2
  Erythrocyte on Day 168 (V4): number analyzed (Participants) | 18
  Erythrocyte on Day 168 (V4): Normal | 17
  Erythrocyte on Day 168 (V4): Abnormal - No clinical significance | 1
  Erythrocyte on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Erythrocyte on Day 336 (V6/EOS): Normal | 25
  Erythrocyte on Day 336 (V6/EOS): Abnormal - No clinical significance | 2
  Protein at Screening (V1): Normal | 24
  Protein at Screening (V1): Abnormal - No clinical significance | 6
  Protein on Day 168 (V4): number analyzed (Participants) | 18
  Protein on Day 168 (V4): Normal | 17
  Protein on Day 168 (V4): Abnormal - No clinical significance | 1
  Protein on Day 336 (V6/EOS): number analyzed (Participants) | 27
  Protein on Day 336 (V6/EOS): Normal | 23
  Protein on Day 336 (V6/EOS): Abnormal - No clinical significance | 4

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | LMIS 50 mg
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMIS 50 mg (N=30)
Perforated ulcer (General disorders) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMIS 50 mg (N=30)
Fatigue (General disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information from the trial is property of the Sponsor and the PI has no right on it except the prior writing authorization of the sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT02712320/SAP_000.pdf
  • Study Protocol (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02712320/Prot_001.pdf